CLINICAL TRIAL: NCT04668755
Title: Effect Of Charcot Restraint Orthotic Walker Three-Dimensional Printed Sole On Charcot Foot Ulcer
Brief Title: Effect of CROW 3d Printed Sole on Charcot Foot Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Haitham Amin Elessawy, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/002367
Record Dates: First submitted 2020-12-05; First posted 2020-12-16 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Charcot Joint of Foot

STUDY DESIGN:
Intervention Model Description: * Sixty patients with Charcot neuroarthropathic foot ulcer (Chronic stage) recruited in the study.
  * Patients divided in to two equal groups in number:
    * Group A (Study group):
  This group compose of 30 patients whom they received the same standard medical treatment as group B in addition fitting with Charcot Restraint Orthotic Walker 3d printed sole for 12 weeks.
  - Group B (Control group): This group compose of 30 patients whom they received the standard medical treatment in addition fitting with Generic Charcot Restraint Orthotic Walker for 12 weeks.
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Charcot Restraint Orthotic Walker 3d printed sole (Active Comparator): the group fit with Charcot Restraint Orthotic Walker 3d printed sole for 12 week. the protocol of gait analysis testing starts with a reacclimation period during which the subject walked usual freely walking across the path for a duration of four minutes and then the testing session data collection done by four acceptable force platform strikes for the feet fitted with the CROW.
  Interventions: Device: Charcot Restraint Orthotic Walker 3d printed sole
- Generic Charcot Restraint orthotic walker (Active Comparator): the group fit with Generic Charcot Restraint Orthotic Walker for 12 week.the protocol of gait analysis testing starts with a reacclimation period during which the subject walked usual freely walking across the path for a duration of four minutes and then the testing session data collection done by four acceptable force platform strikes for the feet fitted with the CROW.
  Interventions: Device: Generic Charcot Restraint orthotic walker

INTERVENTIONS:
Device: Charcot Restraint Orthotic Walker 3d printed sole — The Charcot Restraint Orthotic Walker (CROW) consists of anterior and posterior shells creating a total contact environment based on a rocker sole. the sole is manufactured by 3d printed Metamaterial .
  Manufacture of the 3d printed sole of the CROW paths through two stages ;Computer aided designing (CAD) and computer aided manufacturing (CAM) .
  Arms: Charcot Restraint Orthotic Walker 3d printed sole
Device: Generic Charcot Restraint orthotic walker — It is a clamshell (two piece) design that provides complete/total contact over the shin, calf and foot. The CROW reduces all motion in the ankle and foot to reduce potential for further injury. It is fully padded on the inside, and the bottom is covered with a material similar to shoe soling. It is not worn with a shoe.
  Arms: Generic Charcot Restraint orthotic walker

SUMMARY:
The purpose of the study is to evaluate the therapeutic effect of the Charcot Restraint Orthotic Walker three-dimensional printed sole on Charcot foot ulcer healing.

DETAILED DESCRIPTION:
Foot ulcerations, Charcot neuroarthropathy, and peripheral arterial disease frequently result in gangrene and lower limb amputation. Consequently, foot disorders are leading causes of hospitalization for persons with peripheral neuropathy. Although not all foot complications can be prevented, dramatic reductions in frequency have been achieved by taking a multidisciplinary approach to patient management, The reduction of pressure to the Charcot foot ulcer is essential to treatment. Proper off-loading and pressure reduction prevents further trauma and promotes healing. This is particularly important in the peripheral neuropathy patient with decreased or absent sensation in the lower extremities. Furthermore, recent studies provide evidence that minor trauma (eg, repetitive stress, shoe pressure) plays a major role in the causal pathway to ulceration.

* Off-loading approaches that deal with Charcot neuroarthropathy will decrease the significant psychological, social and functional impact on individuals.
* The need of this study is developed from the lack of controlled studies that reported the therapeutic effect of Charcot Restraint Orthotic Walker 3d printed sole on Charcot foot ulcer.
* So the present study is designed to evaluate the Charcot Restraint Orthotic Walker 3d printed sole on Charcot foot ulcer. Furthermore, the current study may help physical therapist, physicians, and clinicians to organize a protocol of treatment that would be safe, simple and economic for treating patients with Charcot neuroarthropathy.

ELIGIBILITY:
Inclusion Criteria:

* The subject selection will be according to the following criteria: • The patient's ages will range from 45 to 65 years.

  * Both sexes will be included in the study.
  * Informed consent for participation in this study will be obtained in writing from all patients.

Exclusion Criteria:

* The potential participants will be excluded if they meet one of the following criteria:
* Preceding surgical procedure on affected foot.
* Patients on hemodialysis.
* Patients who had any pathological conditions which may affect the results of the study as active malignancy, osteomyelitis and pes planus.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-05 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Force platform to measure peak vertical ground reaction plantar force | Pre-intervention
  Plantar vertical ground reaction force obtained at a rate of 100 Hz measured by Nintendo Wii Balance Board (WBB Nintendo Co. Ltd. Kyoto, Japan) through a four strain gauge sensors (uniaxial vertical force transducers) located at the corners of the board with a usable size of 45 x 26.5 cm were used for data collection; wirelessly via Bluetooth by using third party software illustrates the peak vertical force parameter.
Force platform to measure peak vertical ground reaction plantar force | Three months post-intervention
  Plantar vertical ground reaction force obtained at a rate of 100 Hz measured by Nintendo Wii Balance Board WBB (Nintendo Co. Ltd. Kyoto, Japan) through a four strain gauge sensors (uniaxial vertical force transducers) located at the corners of the board with a usable size of 45 x 26.5 cm were used for data collection; wirelessly via Bluetooth by using third party software illustrates the peak vertical force parameter

SECONDARY OUTCOMES:
Wound Surface area using ImageJ software | Pre-intervention
  The patient is positioned in a comfortable position with exposure of the wound. A ruler as a reference is place directly flat and attach to the skin around the wound area. A photographs were taken including the reference ruler in the images that is captured for the whole wound margins taking in consideration standardization the same angle of capture in the flat mid foot ulcers, but in case of ulcers extend to foot edge, a sterilized transparent grid film (1x1 cm) attached flat on the ulcer then wound margins traced on the transparent grid film and then photographed, then the captured photographs is exported to the computer to be visualized with ImageJ 1.52t software. Surface area measurement of wound margins are traced by the same investigator to establish reliability of measurements
Wound Surface area using ImageJ software | Three months post-intervention
  The patient is positioned in a comfortable position with exposure of the wound. A ruler as a reference is place directly flat and attach to the skin around the wound area. A photographs were taken including the reference ruler in the images that is captured for the whole wound margins taking in consideration standardization the same angle of capture in the flat mid foot ulcers, but in case of ulcers extend to foot edge, a sterilized transparent grid film (1x1 cm) attached flat on the ulcer then wound margins traced on the transparent grid film and then photographed, then the captured photographs is exported to the computer to be visualized with ImageJ 1.52t software. Surface area measurement of wound margins are traced by the same investigator to establish reliability of measurements

CONTACTS AND LOCATIONS:
Overall Officials: Amal M Abd El Baky, PhD, Study Director — faculty of physical therapy
Locations (1):
- Abou Quir General Hospital, Alexandria, Egypt